CLINICAL TRIAL: NCT02470637
Title: A Randomized, Controlled, 6-treatment, 6-sequence, 6-period Cross-over Dose Response Study of 3 Single Doses of Afrezza Inhaled Technosphere Insulin and of 3 Single Doses of SC Insulin Lispro in Patients With Diabetes Mellitus Type 1 Using the Euglycemic Clamp Technique
Brief Title: Single Dose Clamp Study to Evaluate Concentration-time Profile and Metabolic Activity of 3 Dose Levels of Afrezza and 3 Dose Levels of Insulin Lispro in Patients With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PDY14324; 2015-000231-33 (EudraCT Number); U1111-1166-5431 (Other: UTN)
Record Dates: First submitted 2015-06-10; First posted 2015-06-12 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SAR439065 + insulin lispro (Experimental): 1 of 6 sequences with single administration of 3 dose levels of SAR439065 (Afrezza Technosphere insulin) and 3 dose levels of insulin lispro with a washout duration between dosing days (7 to 28 days)
  Interventions: Drug: SAR439065; Drug: Insulin lispro

INTERVENTIONS:
Drug: SAR439065 — Pharmaceutical form:dry powder insulin
  Route of administration: inhalation
  Other Names: Afrezza Technosphere insulin
Drug: Insulin lispro — Pharmaceutical form:solution for injection
  Route of administration: subcutaneous
  Other Names: Humalog

SUMMARY:
Primary Objective:

To assess the dose-response pattern of the glucose consumption (GIR-AUC0-end) of 3 different single doses of Afrezza inhaled Technosphere insulin and of 3 single doses of subcutaneous (SC) insulin lispro in a euglycemic clamp setting.

Secondary Objectives:

To assess the dose proportionality of insulin exposure (INS-AUClast) of 3 different single doses of Afrezza inhaled Technosphere insulin and of 3 single doses of SC insulin lispro in a euglycemic clamp setting.

To assess the pharmacodynamic (PD) characteristics of 3 different single doses of Afrezza inhaled Technosphere insulin and of 3 single doses of SC insulin lispro in a euglycemic clamp setting.

To assess the pharmacokinetic (PK) characteristics of 3 different single doses of Afrezza inhaled Technosphere insulin and of 3 single doses of SC insulin lispro in a euglycemic clamp setting.

To assess the safety and tolerability of 3 different single doses of Afrezza inhaled Technosphere insulin.

DETAILED DESCRIPTION:
The total study duration for one patient is approximately 6.7 to 22.7 weeks (minimum to maximum duration, excluding screening). The duration of the study includes a screening period of 3 to 28 days (D -28 to D -3), 6 treatment periods of 1 or 2 days each (1 overnight stay), a washout period of 7 to 28 days (preferentially 7 days between consecutive dosing), and an end-of-study visit of 7 to 14 days after the last study drug administration.

ELIGIBILITY:
Inclusion criteria :

* Male or female patients, between 18 and 65 years of age, inclusive, with diabetes mellitus type 1 for more than one year, as defined by the American Diabetes Association.
* Total insulin dose of <1.0 U/kg/day.
* Body weight between 50.0 and 95 kg, inclusive, body mass index between 18.5 and 29 kg/m², inclusive.
* Fasting serum C-peptide <0.3 nmol/L.
* Glycohemoglobin (HbA1c) ≤75 mmol/mol (≤9%).
* Stable insulin regimen for at least 2 months prior to study (with respect to safety of the patient and scientific integrity of the study).
* Certified as otherwise healthy for type 1 diabetes mellitus patient by assessment of medical history and physical examination (cardiovascular system, chest and lungs, thyroid, abdomen, nervous system, skin and mucosae, and musculoskeletal system), unless the Investigator considers any abnormality to be clinically irrelevant and not interfering with the conduct of the study (with respect to safety of the subject and scientific integrity of the study).
* Having given written informed consent prior to undertaking any study-related procedure.
* Non-smoking at least for the last 6 months before screening (to be confirmed by urine cotinine <500 µg/L).
* Pulmonary function test at screening: forced expiratory volume in 1 second (FEV1) and forced vital capacity (FVC) >70% of the individual prediction according to the equation of the Third National Health and Nutrition Examination Survey (NHANES III).

Exclusion criteria:

* Severe hypoglycemia resulting in coma/seizures or requiring assistance of another person, and/or hospitalization for diabetic ketoacidosis in the last 6 months before screening visit.
* Frequent severe headaches and/or migraine, recurrent nausea and/or vomiting (more than twice a month).
* Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician.
* History or presence of drug or alcohol abuse (alcohol consumption more than 40 g per day).
* If female, pregnancy (defined as positive beta-human chorionic gonadotropin [β-hCG] blood test), breastfeeding at screening and before any treatment periods (defined as positive β-hCG urine test).
* Any medication (including St John's Wort) within 14 days before inclusion or within 5 times the elimination half-life or PD half-life of the medication, with the exception of insulins, thyroid hormones, lipid-lowering, and antihypertensive drugs and if female with the exception of hormonal contraception or menopausal hormone replacement therapy; any vaccination within 28 days before inclusion.
* Presence or history of any acute or chronic obstructive bronchopulmonary disease including chronic obstructive pulmonary disease, asthma, and cancer.
* Upper respiratory tract infection within 8 weeks before screening.
* Known hypersensitivity to insulin lispro or Afrezza Technosphere insulin and excipients.
* Inability, in the opinion of the Principal Investigator or a designee, to adequately inhale Afrezza powder.
* Any history or presence of deep leg vein thrombosis or a frequent appearance of deep leg vein thrombosis in first-degree relatives (parents, siblings, or children).
* The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Assessment of PD parameter: Area under the glucose infusion rate curve within 24 hours after administration of the investigational medicinal product or until administration of rescue insulin (GIR-AUC0-end) | 24 hours

SECONDARY OUTCOMES:
Assessment of PD parameters: Maximum smoothed glucose infusion rate (GIRmax) | 24 hours
Assessment of PD parameters: Time to GIRmax (GIR-Tmax) | 24 hours
Duration of blood glucose control (time to elevation of smoothed blood glucose profile above different prespecified clamp levels) | 24 hours
Assessment of PK parameters: Area under the baseline-corrected serum insulin concentration-time curve over 24 hours or until administration of rescue insulin (INS-AUClast) | 24 hours
Assessment of PK parameters: Baseline-corrected maximum serum concentration (INS-Cmax) | 24 hours
Assessment of PK parameters: Time to INS-Cmax (INS-Tmax) | 24 hours
Assessment of PK parameters: Area under the concentration-time curve (INS-AUClast) | 24 hours
Number of patients with adverse events | Up to 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 276001, Neuss, Germany

REFERENCES:
- [Derived] Grant M, Heise T, Baughman R. Comparison of Pharmacokinetics and Pharmacodynamics of Inhaled Technosphere Insulin and Subcutaneous Insulin Lispro in the Treatment of Type 1 Diabetes Mellitus. Clin Pharmacokinet. 2022 Mar;61(3):413-422. doi: 10.1007/s40262-021-01084-0. Epub 2021 Nov 13. PMID 34773608